CLINICAL TRIAL: NCT03498053
Title: Smoking Topography Study 2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL63420.068.17
Record Dates: First submitted 2018-01-10; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-03

CONDITIONS: Cigarette Smoking; Smoking Behavior; Cigarette Smoking Toxicity
MeSH Terms: conditions — Cigarette Smoking; Smoking

STUDY DESIGN:
Intervention Model Description: Not-randomized crossover study with a single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cigarette brands smoked by participant (Other): The 3 experimental days per participant are exactly the same, except the cigarette brand they smoke.
  The content of an experimental day is described in the study design.
  Interventions: Behavioral: Marlboro; Behavioral: Marlboro Prime; Behavioral: Marlboro Prime (ventilation holes taped)

INTERVENTIONS:
Behavioral: Marlboro — Participants smoke Marlboro during the first experimental day, ad libitum.
Behavioral: Marlboro Prime — Participants smoke Marlboro Prime during the second experimental day, ad libitum.
Behavioral: Marlboro Prime (ventilation holes taped) — Participants smoke Marlboro Prime (filter ventilation holes taped) during the third experimental day, ad libitum.

SUMMARY:
Rationale: The World Health Organization Framework Convention on Tobacco Control (WHO FCTC) aims for a regulatory strategy including the regulation of the contents of tobacco products (Article 9). Cigarette smoke includes more than 7000 chemicals which are harmful and cause tobacco-related diseases. In the future, regulation of these harmful cigarette constituents should be based on more chemical classes, as the WHO suggested. However, in order to introduce such class-based regulation, a scientific base is needed to define upper limits of allowed amounts of chemicals (groups) in cigarette smoke emissions and to ensure decreased harmful health effects due to cigarette smoking. To date, the causality between human exposure to specific cigarette smoke compounds and the harmful effects is unknown. The first step in closing the gap in knowledge between cigarette smoke exposure and developing tobacco-related diseases includes a proper determination of human exposure to cigarette smoke chemicals. This includes measuring smoking topography and inhalation. Smoking topography is how the smoker smokes the cigarette (puff volume, duration, flow etc). The goal is to link smoking behavior to smoke exposure, for 2 different cigarette brands. The participants will smoke their 'normal' brand Marlboro (experimental day 1) after which they receive the low TNCO (tar, nicotine and carbon monoxide) Marlboro Prime to smoke at home. A week later the experimental day (day 2) is repeated with this cigarette. On the last experimental day (day 3), the participants will smoke the Prime cigarette while the ventilation holes of this low-TNCO cigarette are taped. Afterwards, the personal smoking profiles of the participants, and thus their individual exposures, will be mimicked in the lab using machine smoking. The observed smoking topography and inhalation parameters together give information about the exposure to smoke toxicants. In addition, this study is also designed to measure biomarkers of exposure in body fluids of smokers, such as nicotine and the most abundant cigarette smoke chemicals and their metabolites.

Objective: We want to find out whether the individual habitudinal smoking topography of a smoker smoking his usual brand, and the changes between cigarettes over the day, can be compared to that of smoking a low-TNCO or high nicotine cigarette (i.e. the Marlboro Prime and Red Sun). In addition, differences in inhalation patterns are investigated. Next to that, the exposure will be connected to the nicotine and carbon monoxide levels in blood and/or urine. Also smoke toxicants (and metabolites) in exhaled air, saliva, urine and blood of smokers are determined.

Study design: This prospective observational study monitors smokers in their habitudinal smoking during the day (for 10 hr) while smoking Marlboro, Marlboro Prime and Marlboro Prime taped cigarette, while during the day bodily fluids are sampled at several time points.

Study population: This population consists of 18 Caucasian, healthy, adult males, aged between 25-34 years old. Participants should be used to smoke Marlboro (red/regular) for at least 3 years with a daily average of 13 to 25 cigarettes (about a package every day).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The participating smokers smoke according to their habitudinal smoking pattern, and are therefore not increasingly exposed to the harmful health effects of cigarette smoking. The invasive part of the study is their stay for 3 days (and 1 night when wanted) in a hotel, and the sampling of blood, saliva, urine and exhaled air.

DETAILED DESCRIPTION:
In 2005, the World Health Organization Framework Convention on Tobacco Control (WHO FCTC) was established with the aim for a regulatory strategy as a response to the globalization of the tobacco epidemic. One of their non-price measures to reduce the demand for tobacco includes article 9: Regulation of the contents of tobacco products . Cigarette product regulation is currently based on tar, nicotine and carbon monoxide (TNCO) levels in cigarette smoke, which are indicated on the package. This is not sufficient, since cigarette smoke includes more than 7000 chemicals. There are aldehydes, VOCs, PAHs, nitrosamines, metals and so much more measured in cigarette, causing tobacco-related diseases .

In the future, regulation of these harmful cigarette constituents should be based on more chemical classes, as the WHO suggested. However, in order to introduce such class-based regulation, a scientific base is needed to define upper limits of allowed amounts of chemicals (groups) in cigarette smoke emissions and to ensure decreased harmful effects due to cigarette smoking. To date, the causality between human exposure to specific cigarette smoke compounds and the harmful effects is unknown. The first step in closing the gap in knowledge between cigarette smoke exposure and developing tobacco-related diseases includes a proper determination of human exposure to cigarette smoke chemicals.

Unfortunately, there is a lack of methodology to determine cigarette smoke exposure in humans .

In a prospective observational pilot study in February 2016, natural human smoking behavior was characterized: Smoking Topography Study 2016 (NL55676.068.15). The smoking topography of every smoked Marlboro cigarette was monitored through the CRESSmicro device, which records the puff length, the puff interval, the puff flow and the puff volume. In this study, the investigators could model the individual smoking profiles per participant by using data of 4 random cigarettes. During modelling, puff volume, duration (and thus also flow) and interpuff interval were taken into account.

Since there were no differences in smoking topography of cigarettes smoked observed at different times of the day implies that in this new study, the researchers can invite participants for a shorter time because only data of 4 cigarettes is needed to adequately model their overall smoking profile needed for exposure measurements. These smoking topography parameters are needed for the settings of a smoking machine, applied to mimic the exact exposure to cigarette smoke toxicants for each individual.

In our previous study the researchers concluded that smokers have their own individual smoking topography. Of course, smoking is also accompanied by the inhalation of harmful chemicals, but the smoker is not aware of this during smoking and therefore does not adapt his smoking topography with respect to that exposure. However, it is unknown by what means the individual smoking topography parameters are related to toxicant exposure in the different parts of the lungs. For example, higher puff volumes with a different composition of toxicants lead to a different inhalation pattern than small puff volumes, possible followed by different exposure in the lungs.

In this new study the researchers want to include respiratory parameters of breathing and inhalation over the day as well. Until now, inhalation risk assessment is based on human breathing patterns, while breathing and inhaling smoke are not the same due to the presence of harsh compounds in the smoke. The current study aims to measure respiratory parameters to identify which lung compartments are exposed to what extent in relation to the observed smoking topography. This can be achieved by respiratory inductive plethysmography (RIP), a non-invasive device that can be worn throughout the day. In the current study, the Hexoskin will be applied for these measurements.

Literature describes that the process of smoking topography and inhalation differs per cigarette and situation . In other words, the smoker doses himself to gain nicotine, with additional production of carbon monoxide (CO) and other harmful cigarette smoke-associated chemicals.

As described before, in the future cigarettes will be changed as they are only allowed to contain a maximum of certain toxicants. One of the options to make cigarettes less addictive is to add less nicotine. It is known that smokers show compensating behavior when smoking other cigarettes than their used to, to gain the same amount of nicotine. Our machine smoking experiments show that when smoking low-TNCO cigarettes, the composition of the smoke per mg nicotine changes under the same smoking conditions. This means that the cigarette characteristics are also at least partly responsible for the smoke composition. The researchers are interested in how smoking behavior and inhalation, and thus exposure, changes when offering a smoker another type of cigarette.

Therefore, the researchers are interested whether the smoking behavior changes when the smoker has to smoke a low TNCO cigarette, i.e. the Marlboro Prime. The low values of nicotine in the smoke of the Marlboro Prime are partly achieved by ventilation holes in the cigarette filter. By closing these filter vents with tape around the filter, the smoke is no longer diluted with side stream air, and the cigarette design is slightly different.

The participants will smoke their 'normal' brand Marlboro (day 1). After the experimental day, they receive the Marlboro Prime for smoking at home, so they get used to smoking a 'new' cigarette. A week later the experimental day (day 2) is repeated with this cigarette. The participants can stay overnight, or come back the next day (day 3) to smoke the Prime cigarette while the ventilation holes of this low-TNCO cigarette are taped. See the scheme in Table 1.

As in the STS2016, this study again is aimed at measuring smoking in a habitual rhythm without imposing it as has been done thus far , , . With this, the natural smoking topography per cigarette can be measured, in combination with the respiratory parameters by wearing a non-invasive RIP device. By providing the participants with the Marlboro Prime cigarettes prior to the experimental days 2 and 3, they can get used to smoking them at home in order to develop 'natural' smoking behavior.

As during the last study, the sampling is following a sampling scheme (Figure 1). In summary, during the day, blood, exhaled air, urine and saliva will be sampled to measure nicotine, carbon monoxide, but also other cigarette smoke compounds, such as aldehydes and their metabolites.

In the future, the personal smoking regimes of the participants, and thus their personal exposures, will be mimicked with machine smoking experiments. This will be linked to the RIP parameters.

Points of attention that came out of the STS 2016, include that smokers smoked less cigarettes than expected. Reason for that is, as they mentioned, that they cannot smoke in the apartment, while they smoke inside at home. Another reason was that they have to smoke alone, while at home or work there often is a co-smoker. The participants didn't experience difficulties or changes in smoking behavior due to the use of CRESS. They all 'practiced' smoking with the CRESS the evening before the experimental day. In the present study 2 smokers will be invited at the same time. Again, smokers have to go outside for a smoke to protect the researchers to secondhand smoke exposure. This is kept as attainable as possible.

Primary Objective:

Is there a difference in natural smoking topography between Marlboro, Marlboro Prime and Marlboro Prime taped leading to a different exposure for the smoker?

Secondary Objective(s):

Is it possible to map personal smoking profiles with only 4 random cigarettes, as showed in the previous Smoking Topography Study 2016?

Is a different smoking topography profile per smoker related to deviating exposure of mainstream smoke in the respiratory tract compartments, for the different cigarettes?

Can exhaled air of smokers be used as biomarker for exposure to VOCs/aldehydes?

Are nicotine and toxicant (metabolite) levels in blood/urine changing over the day and connected to the smoking behavior of the different cigarettes?

Study Design The Smoking Topography Study 2018 is a not-randomized cross-over study with a single group, with the duration of 3 months. Participants will visit our research apartment at Apart Hotel Randwyck, for 1 day in the first week and 2 days in the second week (Table 1).

An experimental day starts at 08.00hr and ends at 19.00hr (Figure 1). The different study days have exactly the same set-up with the cigarette brand smoked during the day being the only difference. In this study it is important that the participants are able to smoke cigarettes 'ad libitum'. Because it is impossible to monitor this smoking topography at home, The smoking topography is measured at a research location. Therefore, this study takes place in an apartment at Hotel Randwyck in a homelike atmosphere where standardized meals are served and cigarettes can be smoked when and how the participant desires. The smoking topography of every smoked cigarette will be monitored through the CRESSmicro device, which records the puff length, the puff interval, the puff flow and the puff volume . Furthermore, the exact time point of smoking (i.e. the moment the cigarette is lit) is noted in the experiment time table.

Due to this setup, the smoking topography measurements do not take place at scheduled time points and therefore only 2 participants per day will be measured. Total duration of the study will be 3 months, including 18 smoking individuals (Table 1).

Participants are their own controls by measuring baseline samples (t=baseline). This sampling takes place upon arrival, before the first cigarette is smoked. Consequently, participants are asked not to smoke when waking up, but to wait upon their arrival at the research location. These baseline samplings include the collection of urine, exhaled air, blood, a mouth swap and saliva.

Goal of a study day is to follow the smoker in his personal daily life smoking schedule. They can smoke when they want or feel the urge to smoke. Therefore, the sampling time points and the amount of cigarettes smoked are unknown per participant (Figure 1). Despite the unknown time points on forehand, smoking topography of every single cigarette within their presence at the research apartment is measured. During the whole experiment, experimental time is used. The start of the experiment (expected to be around 09.00hr) is the start of the experimental day, noted as timepoint 0. This is probably shortly after the baseline measurements.

All spent cigarette butts are collected in separate plastic tubes per participant with the experimental smoking time noted. Because it is very important not to interfere with the daily life smoking schedule, the experiment day is divided into timeslots for urine and a fixed time point for saliva sampling.

Urine will be collected at baseline and during 2 time periods. The first time point includes the baseline measurement before the first cigarette is smoked. Next, all urine between t=0 and t=5 hours is collected in 1 beaker and urine between t=5 and t=10 is collected in another beaker. The participant is asked to empty his bladder just before the timeslots end. This results in 3 urine samples per participant.

Saliva and a mouth swap are collected at t=baseline, t=0 (immediately after the first cigarette), t=5 and t=10. This results in 4 saliva samples and mouth swaps per participant.

The exhaled air and blood samples are collected before and immediately after smoking a cigarette to have the most accurate measure associated with the cigarette smoking. However, the smoking time points are uncertain due to the chosen setup of this study. However, since all smokers included smoke around 20 cigarettes a day, they will at least smoke every 2 to 2.5 hours. Therefore, time periods of 2.5 hours in which the first cigarette smoked is used for sampling blood and exhaled air, immediately after finishing smoking.

At baseline, the participant is asked to exhale via the nosemouth cap of the Owlstone (a breathing device) whereby the exhaled air passes the adsorption tubes. The exhaled air just before and after finishing smoking the first cigarette is collected (t=0). The same is done for cigarettes smoked between t=2.5 and t=5, between t=5 and t=7.5, between t=7.5 and t=10 and the last sampling at T=10. This results in 7 exhaled air samples per participant.

To avoid multiple punctures, the participants get a peripheral venous canula at baseline, after which the baseline blood sample is withdrawn. The next blood sample is withdrawn just before and after finishing smoking the first cigarette (t=0). Then, the sampling points are just before and immediately after the first cigarette between t=0 and t=2.5, between t=2.5 and t=5, between t=5 and t=7.5, between t=7.5 and t=10 and the last sampling is at T=10. For analysis of blood aldehydes an extra blood sample will be drawn from the canula at baseline and immediately after the first cigarette as well as immediately before and after the first cigarette after t=5 and t=7.5. This results in 13 blood sampling points per participant.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 25-35 years old (birth year 1982 - 1992)
* Caucasian
* Smoking Marlboro as usual brand for at least 3 years
* Used to smoke between 13 and 25 cigarettes a day (around a package/day)

Exclusion Criteria:

* Heavy smoker (minimum of 25 cigarettes/day)
* Smokes more than 1 brand on a regular base.
* Amount of cigarettes per day varies ±10, between days
* Daily medication use
* Experienced adverse effects due to smoking
* Suffering chronic illness

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Nicotine metabolism is influenced by the menstrual cycle for females, therefore thy are excluded from the study
Enrollment: 12 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Natural smoking behavior: amount | 3 days
  number of cigarettes
Puffing parameters: volume | 3 days
  puff volume (ml)
Puffing parameter: duration | 3 days
  puff duration(sec)
Puffing parameter: amount | 3 days
  puff number
Puffing parameter: interval | 3 days
  interpuffinterval(sec)

SECONDARY OUTCOMES:
Biomarkers in blood | 13 times in 3 days
  Nicotine, cotinine, aldehyde adducts in blood
Biomarkers in urine | 13 times in 3 days
  Nicotine, cotinine, aldehyde adducts in urine

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Boots, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burns DM, Dybing E, Gray N, Hecht S, Anderson C, Sanner T, O'Connor R, Djordjevic M, Dresler C, Hainaut P, Jarvis M, Opperhuizen A, Straif K. Mandated lowering of toxicants in cigarette smoke: a description of the World Health Organization TobReg proposal. Tob Control. 2008 Apr;17(2):132-41. doi: 10.1136/tc.2007.024158. No abstract available. PMID 18375736
- [Result] Marian C, O'Connor RJ, Djordjevic MV, Rees VW, Hatsukami DK, Shields PG. Reconciling human smoking behavior and machine smoking patterns: implications for understanding smoking behavior and the impact on laboratory studies. Cancer Epidemiol Biomarkers Prev. 2009 Dec;18(12):3305-20. doi: 10.1158/1055-9965.EPI-09-1014. PMID 19959678
- [Result] Wood T, Wewers ME, Groner J, Ahijevych K. Smoke constituent exposure and smoking topography of adolescent daily cigarette smokers. Nicotine Tob Res. 2004 Oct;6(5):853-62. doi: 10.1080/1462220042000282537. PMID 15700921
- [Result] Hammond D, Fong GT, Cummings KM, Hyland A. Smoking topography, brand switching, and nicotine delivery: results from an in vivo study. Cancer Epidemiol Biomarkers Prev. 2005 Jun;14(6):1370-5. doi: 10.1158/1055-9965.EPI-04-0498. PMID 15941943
- See also: WHO Framework Convention on Tobacco Control. ISBN: 9241591013 — http://apps.who.int/iris/bitstream/10665/42811/1/9241591013.pdf